**ID:** Therapeutic Touch And Music

NCT ID not yet assigned

**İntial Release: 21.09.2021** 

Variables of the Study

Dependent Variable: The mean scores obtained from the PSQI, MSDS, and MÖYQÖ scales

constitute the dependent variables of the study.

Independent Variable: Therapeutic Touch and Music Concert practices constitute the

independent variable of the research.

Control Variables: Women's socio-demographic characteristics (age, education level,

occupation, economic status, marital status, family type, body mass index, number of children,

chronic disease status, smoking and alcohol use) and menopausal information (menopausal or

not). absence, menstrual cycle and menopause duration) constituted the control variables of the

study.

**Statistical Analysis of Research Data** 

IBM SPSS Statistics 22.0 package for evaluation of research data program was used. In the

evaluation of the data, percentage, mean, standard deviation, normal distribution, t-test in

independent groups, t-test in dependent groups and ANOVA tests, multiplex linear regression

and correlation analyzes were used. Statistical significance level p;0.05 has been accepted as.